CLINICAL TRIAL: NCT01393197
Title: Clinical Trial of Transcatheter Arterial Chemoembolization (TACE)With KMG Microsphere Treating Advance-stage Hepatocellular Carinomas
Brief Title: Transcatheter Arterial Chemoembolization With KMG Microsphere Treating Advance-stage Hepatocellular Carinomas (TACE-KMG)
Acronym: TACE-KMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TMU-CIH-IR-003
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2010-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TACE -oil (Active Comparator): embolization agent:Iodinated Oil or /and gelatin sponge Iodinated Oil （5-30ml）with Epirubicin （30-40mg/m2） or and gelatin sponge
  Interventions: Other: Therapeutic Chemoembolization
- TACE-KMG ( routine dose Chemo) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g) with routine dose Epirubicin （30-40mg/m2）
  Interventions: Other: Therapeutic Chemoembolization
- TACE-KMG( low dose Chemo ) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g) with low dose Epirubicin （5-10mg/m2）
  Interventions: Other: Therapeutic Chemoembolization
- TACE-KMG(without chemo) (Experimental): embolization agent:KMG microsphere( 150-450µm,0.2-2g)
  Interventions: Other: Therapeutic Chemoembolization

INTERVENTIONS:
Other: Therapeutic Chemoembolization — Transcatheter Arterial Chemoembolization
  Other Names: Transcatheter Arterial Chemoembolization，TACE

SUMMARY:
The purpose of this study is to evaluate the effects of Transcatheter Arterial Chemoembolization (TACE) with KMG microsphere in treating HCC. And to determine which one is better,KMG microsphere or lipiodol?

DETAILED DESCRIPTION:
The most important part of effect in TACE is embolization .But there is no clinical trials on which one is better,KMG microsphere or lipiodol? what effect did chemo play in the TACE treating HCC? Which one is better,routine dose or low dose? Experts in USA and Japan had their own researches and standpoints.We think it is important to push a clinical trail to answer these problem.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular Carinomas with diagnosis of pathology or cytology or consistent with China 2001 guideline of Clinical Diagnosis Hepatocellular Carinomas clinical stage（The Barcelona Liver Clinic staging system,BCLC B and C)，or can not receive surgical intervention
* liver function:Child-Pugh A、B
* PST 0-1（Eastern Cooperative Oncology Group Performance Score ,ECOG）
* Lifespan≥6 months
* First time to receive treatment
* Can accept the follow up
* informed consent was gotten
* the number of lesion ≤ 5

Exclusion Criteria:

* pregnant or lactation woman
* emotional disturbance
* serious heart ,lung disfunction or serious diabetes mellitus
* serious reactiveness infections;（exp:type B or C hepatitis）
* liver function :Child-Pugh Score C
* thrombocyte<6×109/L
* diffuse HCC
* widespread metastasis
* serious atherosclerosis
* acquired immunodeficiency syndrome;AIDS
* thrombosis or thrombosis event in 6 months
* renal inadequacy who need hemodialysis or peritoneal dialysis
* with other tumors except basal cell carcinoma and carcinoma in situ of cervix
* serious alimentary tract hemorrhage in 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2480 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 3 years
  Time to progression

SECONDARY OUTCOMES:
total survival | 3 years
  total survival
remission rate | 3 years
  remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Guo, MD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- See also: Related Info — http://www.tjmuch.com/